CLINICAL TRIAL: NCT02154698
Title: A Multi-center Study Comparing Standard 22-gauge and 22-gauge ProCore Needles for Endobronchial Ultrasound
Brief Title: 22-gauge ProCore Needle v. Standard 22-gauge (P00030500)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Cook Endoscopy (Industry); University of North Carolina (Other); Johns Hopkins University (Other); Thoraxklinik-Heidelberg gGmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 00030500
Record Dates: First submitted 2014-05-22; First posted 2014-06-03 (Estimated); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Quantity of Tissue Obtained; Quality of Tissue Obtained; Ease of Use of 22-gauge ProCore EBUS Needles and the Standard 22-gauge Needles

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 22-gauge Standard Needle (Active Comparator): Participants will have each node sampled starting with the standard 22G needle on the first pass followed by the ProCore 22G needle on the second pass (for a total of 8 passes)
  Interventions: Other: 22-gauge Standard Needle
- 22-gauge ProCore Needle (Active Comparator): Participants will have each node sampled starting with the ProCore 22G on the first pass followed by the standard 22G needle on the second pass (for a total of 8 passes)
  Interventions: Other: 22-gauge ProCore Needle

INTERVENTIONS:
Other: 22-gauge Standard Needle — Acquisition of lymph nodes samples using the 22-gauge Standard Needle, following subject-sedation and the introduction of an EBUS scope into the airway.
  Arms: 22-gauge Standard Needle
Other: 22-gauge ProCore Needle — Acquisition of lymph nodes samples using the 22-gauge ProCore Needle, following subject-sedation and the introduction of an EBUS scope into the airway.
  Arms: 22-gauge ProCore Needle

SUMMARY:
The purpose of this study is to compare the usefulness of two needles (used for obtaining a lung tissue sample : (1) standard 22-gauge, and (2) ProCore 22-gauge) for endobronchial ultrasound

DETAILED DESCRIPTION:
The purpose of this study is to compare the usefulness of two needles used for obtaining a lung tissue sample: (1) standard 22-gauge, and (2) ProCore 22-gauge. Both of these needles are used to get biopsies (samples) of lung tissue. The standard needle has one bevel (angled side of the needle formed when it is sharpened to make a point), while the ProCore needle has 2 bevels. The standard needle is more commonly used and we are doing this study to see if the ProCore needle would be more useful.

The investigator in charge of this study is Dr. Nichole T. Tanner. This study is being done at four sites and will involve approximately 200 volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with known or suspected lung cancer with mediastinal adenopathy as defined by a mediastinal lymph node >1 cm in short axis or a normal sized lymph node with uptake on FDG-PET scan that is higher than background PET activity.
2. Participants must be at least 18 years old or older, lack bleeding disorders, and be able to provide informed consent. The latter two criteria will be assessed from the patient's history and the consenting interview.

Exclusion Criteria:

1. Subjects who refuse to participate, or demonstrate inability to give informed consent
2. Subjects who are less than 18 years of age
3. Subjects who lack fitness for flexible bronchoscopy as determined by the physician performing the bronchoscopy before the procedure
4. Subjects with suspected sarcoidosis, lymphoma, or metastatic cancer from other sites (i.e. those without a known or suspected lung primary)
5. Subjects on anticoagulation (other than Aspirin) whom cannot have their anticoagulation held for the procedure due to other clinical reasons (i.e. recent cardiac stent placement).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2017-12-19 (Actual); Study Completion 2017-12-19 (Actual)

PRIMARY OUTCOMES:
Ease of use of 22-gauge ProCore EBUS needles and the standard 22-gauge needles. | Within two weeks from the day of the procedure
Quality of tumor obtained (measured by cell block and ability to perform mutational analysis) | Within two weeks from the day of the procedure
Quantity of tissue obtained (measured by number of unstructured fragments) | Within two weeks from the day of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Nichole T Tanner, MD, M.S.C.R, Principal Investigator — Medical University of South Carolina
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - University of North Carolina Medical School, Chapel Hill, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina